CLINICAL TRIAL: NCT05141851
Title: The Impact of Thread Length on Implant Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Responsible Party: Principal Investigator, Vanessa Rocha Rodrigues, Vanessa Rocha Rodrigues, University of Lisbon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The impact of thread length on
Record Dates: First submitted 2021-11-20; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Implant Stability
Keywords: implant stability; implant threads

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implants with 0,7mm threads (Active Comparator): Placement of Implants with 0,7mm threads
  Interventions: Device: Implants with 0,7 mm threads
- Implants with 0,3mm threads (Active Comparator): Placement of Implants with 0,3mm threads
  Interventions: Device: Implants with 0.3 mm threads

INTERVENTIONS:
Device: Implants with 0,7 mm threads — Implants were placed, with threads of 0.7 mm in the location of premolars and molars.
  Arms: Implants with 0,7mm threads
Device: Implants with 0.3 mm threads — Implants were placed, with threads of 0.3 mm in the location of premolars and molars.
  Arms: Implants with 0,3mm threads

SUMMARY:
Some studies show that different types of threads in tapered implants result in differences in primary stability. The aim of this study is to a perform a prospective, controlled, randomized clinical trial comparing primary and secondary stability between long and standard thread implants in the treatment of partial edentulous patients.

DETAILED DESCRIPTION:
The study sample consists of 23 maxillary partial edentulous patients, where 32 implants were placed, with threads of 0.7 mm or 0.3 mm in the location of premolars and molars. The comparison, in terms of primary stability, is made by measuring the ISQ value (implant stability quotient), in four locations (buccal, palatal, mesial and distal). Statistical analysis was performed using the independent T-Test.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 18 years;
* No systemic conditions that contraindicate surgery;
* Periodontal health or periodontal disease treated as part of a periodontal support program and having a high level of plaque control;
* Partial edentulous patients, in the upper jaw, specifically in the location of premolars and molars;

Exclusion Criteria:

* Patients with insufficient quantity of bone for implant placement without bone regeneration procedures;
* Patients who underwent medication that could affect stability and osteointegration up to 3 months prior to study initiation;
* Patients with untreated periodontal pathology or who have not followed periodontal supportive treatment;
* Smokers, Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
primary dental implant stability | On the 1 day of implants placement
  measuring the ISQ value (implant stability quotient)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Mascarenhas, PhD, Study Director — University of Lisbon; Susana Noronha, PhD, Study Director — University of Lisbon; Vanessa Rodrigues, Dr, Principal Investigator — University of Lisbon
Locations (1):
- Vanessa Rodirgues, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No